CLINICAL TRIAL: NCT02473302
Title: Preventive Strategies in Colorectal Carcinogenesis Production and Meat Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government)
Responsible Party: Principal Investigator, Adeline BLOT, Clinical research assistant, University Hospital, Clermont-Ferrand
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Securiviande
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — ATF7IP protein, human; Tocopherols

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- ham (Placebo Comparator): 160g per day during 4 days
  Interventions: Other: ham
- ham + pomegranate extract (Experimental): 160g per day during 4 days
  Interventions: Other: ham + pomegranate extract
- ham + tocopherol (Experimental): 160g per day during 4 days
  Interventions: Other: ham + tocopherol
- rare sirloin steak (Placebo Comparator): 110g per day during 4 days
  Interventions: Other: rare sirloin steak
- marinated rare sirloin steak (Experimental): 110g per day during 4 days
  Interventions: Other: marinated rare sirloin steak
- marinated cooked sirloin steak (Experimental): 110g per day during 4 days
  Interventions: Other: marinated cooked sirloin steak

INTERVENTIONS:
Other: ham — 160g per day during 4 days
  Arms: ham
Other: ham + pomegranate extract — 160g per day during 4 days
  Arms: ham + pomegranate extract
Other: ham + tocopherol — 160g per day during 4 days
  Arms: ham + tocopherol
Other: rare sirloin steak — 110g per day during 4 days
  Arms: rare sirloin steak
Other: marinated rare sirloin steak — 110g per day during 4 days
  Arms: marinated rare sirloin steak
Other: marinated cooked sirloin steak — 110g per day during 4 days
  Arms: marinated cooked sirloin steak

SUMMARY:
Colorectal Cancer is, in non-smokers for both sex, first cause of cancers mortality in Western country.

The main risk factors associated with colorectal cancer depend of lifestyle, and processed meat and red meat could be involved in carcinogenesis by cytotoxic and genotoxic compound linked to lipid peroxidation and nitrosation.

The aim of this study is to study the impact of the daily consumption of beef, processed or not, on lipid peroxidation induced heme iron ; and to study the impact of the daily consumption of ham, processed or not, on the nitrosilation induced heme iron.

DETAILED DESCRIPTION:
24 healthy volunteers will be randomized and will start the study. The study will last 12 weeks for each subject. The first week will be a week of adaptation (or run-in period) to the diet which they will have to follow for the duration of study. During this period, they will collect 3 samples of stools and urine. Then subjects will alternate 4 days of diet either with ham, or with ham and pomegranate extract, or with ham enriched with vitamin E or sirloin steak, marinated sirloin steak or marinated cooked sirloin steak. At least, 3 days will separate every period (wash-out) of nutritional intervention. Urines and stools will be collected last 3 days of every interventional period and also last day of every wash out period.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Body mass index 20 <= BMI <= 30 kg/m2
* Affiliated to French National Health Insurance
* Subject giving his written informed consent
* Subject considered as normal after clinical examination and medical questionnaire

Exclusion Criteria:

* Previous medical and/or surgery judged by the investigator as incompatible with this study
* Previous familial of colon, ovarian or breast cancer
* Chronic pathologies : cardiovascular diseases, cancer, chronic inflammation diseases, renal, intestinal impairments
* Dislike ham or red meat
* Heavy consumer of alcohol
* Practising intensive physical exercise (> 5 hours)
* Being under someone's supervision
* Refusal to be registered on the National Volunteers Data file
* Dietary habits unreliable to controlled food intake
* Being in exclusion on the National Volunteers Data file

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Fecal marker | 12 weeks
  TBARS Fecal for red meat pane and NOCs Fecal for ham

SECONDARY OUTCOMES:
NOC | 12 weeks
  Fecal marker for red meat pane
cytotoxic activity of fecal water | 12 weeks
  Fecal marker for red meat pane
DHN-MA | 12 weeks
  urinary marker for red meat pane
TBARs | 12 weeks
  Fecal marker for ham
cytotoxic activity of fecal water | 12 weeks
  Fecal marker for ham
DHN-MA | 12 weeks
  urinary marker for ham

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice PIERRE, Phd, Study Chair — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement; Noel CANO, Md, Phd, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CRNH Auvergne, Clermont-Ferrand, Auvergne, France